CLINICAL TRIAL: NCT01432015
Title: A Phase IV Study Comparing the Efficacy of Fosaprepitant to Aprepitant for Chemotherapy Induced Nausea and Vomiting in Patients Treated for Gynecological Cancer
Brief Title: Fosaprepitant Versus Aprepitant in the Prevention of Chemotherapy Induced Nausea and Vomiting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gynecologic Oncology Associates (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GOA-NVM1
Record Dates: First submitted 2011-09-07; First posted 2011-09-12 (Estimated); Results first posted 2015-05-27 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2015-05

CONDITIONS: Ovarian Cancer; Uterine Cancer
Keywords: aprepitant; fosaprepitant; gynecologic cancer; emesis
MeSH Terms: conditions — Ovarian Neoplasms; Uterine Neoplasms; Vomiting | interventions — fosaprepitant; Aprepitant; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fosaprepitant (Active Comparator): Fosaprepitant for Injection 150 mg is administered intravenously on Day 1 only as an infusion over 20-30 minutes initiated approximately 30 minutes prior to chemotherapy. Oral Placebo given on days 1-3
  Interventions: Drug: fosaprepitant; Other: Oral Placebo
- Aprepitant (Active Comparator): Aprepitant 125 mg orally 1 hour prior to chemotherapy treatment (Day 1) and 80 mg orally once daily in the morning on Days 2 and 3. 100 cc of IV placebo administered on day 1
  Interventions: Drug: aprepitant; Other: IV placebo

INTERVENTIONS:
Drug: fosaprepitant — Fosaprepitant for Injection 150 mg is administered intravenously on Day 1 only as an infusion over 20-30 minutes initiated approximately 30 minutes prior to chemotherapy. Patient will receive standard pre-medications
  Other Names: Emend IV
  Arms: Fosaprepitant
Drug: aprepitant — Aprepitant 125 mg orally 1 hour prior to chemotherapy treatment (Day 1) and 80 mg orally once daily in the morning on Days 2 and 3. patient will receive standard pre-medications
  Other Names: Emend
  Arms: Aprepitant
Other: Oral Placebo — One pill administered on days 1-3 in conjunction with Fosaprepitant.
  Arms: Fosaprepitant
Other: IV placebo — 100 cc of IV placebo administered on day in conjunction with Aprepitant
  Other Names: Normal Saline
  Arms: Aprepitant

SUMMARY:
Nausea and vomiting are two of the more concerning adverse outcomes associated with chemotherapy in the treatment of gynecologic malignancies. In fact, nearly 90% of cancer patients develop chemotherapy induced nausea and vomiting (CINV) following treatment with carboplatin and paclitaxel. The successful control of chemotherapy induced nausea and vomiting (CINV) is thus, of paramount importance in ensuring optimal treatment and sustaining a cancer patient's quality of life.

DETAILED DESCRIPTION:
Studies have indicated that oral and intravenous anti-emetics are equivalent with regard to efficacy; when evaluating cost and convenience, the intravenous route may be preferable. Fosaprepitant, a water-soluble phosphoryl prodrug for aprepitant, is converted to aprepitant via phosphatases following intravenous administration. Given the rapid conversion of fosaprepitant to the active form (i.e., aprepitant), the two medications appear to provide a similarly effective antiemetic impact. Clinical reports have additionally suggested that fosaprepitant could be appropriate as an intravenous alternative to the oral aprepitant.

ELIGIBILITY:
Inclusion Criteria:

* Female Gender
* Age > 18 years
* A histologic diagnosis of stage III/IV gynecologic cancer (e.g., epithelial ovarian, fallopian tube, peritoneal cancer and uterine cancer).
* Subjects who will be treated with Taxol and Carboplatin as standard of care for a newly diagnosed gynecological cancer.
* Adequate bone marrow function as demonstrated by:

Absolute neutrophil count (ANC) > 1,500/μL; platelet count > 100,000/μL; and hemoglobin > 9 g/dL • Adequate renal function demonstrated by: Serum creatinine of < 1.5 x ULN or 24-hr measured urine creatinine clearance > 60 mL/min for patients with serum creatinine > 1.5 x ULN

• Adequate hepatic function demonstrated by: Total bilirubin of < 1.5 x ULN AST or ALT ≤ 2.5 x ULN

* EGOG status of < 2: Postoperatively, patients demonstrate an ECOG score of 1 or 2. However, during the first cycle of chemotherapy, the patients' performance status improves to < 1.
* Projected life expectancy of at least 3 months
* Ability to comply with the visit schedule and assessments required by the protocol
* Negative pregnancy test for women of childbearing potential
* Signed, IRB approved informed consent and HIPPA consent

Exclusion Criteria:

* Subjects with a diagnosis of epithelial ovarian, fallopian tube or peritoneal cancers of low malignant potential (borderline carcinomas) are not eligible.
* Allergy or intolerance to 5HT3 or NK-1 antagonists and dexamethasone
* An episode of vomiting or retching within 24 hours before the start of the initial treatment with chemotherapy
* Subjects with concomitant malignancy or a previous malignancy within the past three (3) years (except non-melanoma skin cancer)
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study.
* Screening clinical laboratory values of:

ANC of <1500/DL Platelet count of <100,000/µL Total bilirubin of *1.5 mg/dL x ULN SGOT (AST) or SGPT (ALT) * 2.5 x ULN Serum creatinine of * 1.5 mg/dL Hemoglobin of * 9 gm/dL (may be transfused or receive a colony stimulating factor to maintain or exceed this level)

* EGOG status of > 2
* Gastrointestinal obstruction or an active peptic ulcer
* Patients who are pregnant or breast feeding because aprepitant may be harmful to the developing fetus and newborn
* Known active HIV and viral hepatitis infections
* Inability to comply with study
* New York Heart Association (NYHA) Grade II or greater congestive heart failure (see Appendix D)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John P Micha, MD, Principal Investigator — Gynecologic Oncology Associates
Locations (1):
- Gynecologic Oncology Associates, Newport Beach, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Fosaprepitant and Placebo: Fosaprepitant for Injection 150 mg is administered intravenously on Day 1 only as an infusion over 20-30 minutes initiated approximately 30 minutes prior to chemotherapy.Oral Placebo 125 mg given 1 hour prior to infusion of chemotherapy on day 1 and oral Placebo 80 mg on day 2 and day 3. Patient will receive standard pre-medications on day 1
- Aprepitant and Placebo: Aprepitant is 125 mg orally 1 hour prior to chemotherapy treatment (Day 1) with Intravenous Placebo on day 1 and 80 mg orally once daily in the morning on Days 2 and 3. patient will receive standard pre-medications on day 1.
Period: Overall Study
Arm/Group | Fosaprepitant and Placebo | Aprepitant and Placebo
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Fosaprepitant Including Placebo: Fosaprepitant (EMEND™) for Injection 150 mg is administered intravenously on Day 1 only as an infusion over 20-30 minutes initiated approximately 30 minutes prior to chemotherapy.Oral Placebo 125 mg given 1 hour prior to infusion of chemotherapy on day 1 and oral Placebo 80 mg on day 2 and day 3.Patient will receive standard pre-medications on day 1
  Aprepitant (EMEND™) is 125 mg orally 1 hour prior to chemotherapy treatment (Day 1) and 80 mg orally once daily in the morning on Days 2 and 3
  fosaprepitant including placebo: Fosaprepitant for Injection 150 mg is administered intravenously on Day 1 only as an infusion over 20-30 minutes initiated approximately 30 minutes prior to chemotherapy. Patient will receive standard pre-medications
- Aprepitant Including Placebo: Aprepitant (EMEND™) is 125 mg orally 1 hour prior to chemotherapy treatment (Day 1) with Intravenous Placebo and 80 mg orally once daily in the morning on Days 2 and 3 with Placebo Intravenously on day 1. patient will receive standard pre-medications on day 1.
  aprepitant including placebo: Aprepitant 125 mg orally 1 hour prior to chemotherapy treatment (Day 1) and 80 mg orally once daily in the morning on Days 2 and 3. patient will receive standard pre-medications
- Total: Total of all reporting groups
Arm/Group | Fosaprepitant Including Placebo | Aprepitant Including Placebo | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 9 | 17
  >=65 years | 2 | 1 | 3
Sex/Gender, Customized [Number; unit: participants]
  Female | 10 | 10 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 9 | 10 | 19
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Secondary Outcome: Impact on Daily Living Activities
Description: Proportion of patients reporting no impact on daily living activities following initiation of chemotherapy
Time Frame: 13 months
Population: Study participants included adult, female patients with a histologically confirmed, newly diagnosed gynecologic cancer (e.g., epithelial ovarian, fallopian tube, primary peritoneal cancer or uterine cancer).
Measure: Number; unit: percentage of participants
Arm/Group | Fosaprepitant Including Placebo | Aprepitant Including Placebo
Number analyzed (Participants) | 10 | 10
percentage of participants | 10 | 10

2. Primary Outcome: Overall Complete Response Rate
Description: no emetic episodes or rescue therapy following the initiation of chemotherapy
Time Frame: 13 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Fosaprepitant Including Placebo | Aprepitant Including Placebo
Number analyzed (Participants) | 10 | 10
percentage of participants | 10 | 10

ADVERSE EVENTS:
Time Frame: The adverse events were reviewed and collected 28 days after treatment
Groups:
- Fosaprepitant and Placebo: Fosaprepitant for Injection 150 mg is administered intravenously on Day 1 only as an infusion over 20-30 minutes initiated approximately 30 minutes prior to chemotherapy.Oral Placebo 125 mg given 1 hour prior to infusion of chemotherapy on day 1 and oral Placebo 80 mg on day 2 and day 3.Patient will receive standard pre-medications on day 1
Arm/Group | Fosaprepitant and Placebo | Aprepitant and Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No